CLINICAL TRIAL: NCT03793036
Title: A Randomized Controlled Study of Preoperative Oral Carbohydrate Loading Versus Fasting in Patients Undergoing Colorectal Surgery
Brief Title: Preoperative Administration of Oral Carbohydrate Drink and Postoperative Insulin Resistance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nermina Rizvanović (Other)
Responsible Party: Sponsor-Investigator, Nermina Rizvanović, MD Anesthesiology and Intensive Care Specialist, Cantonal Hospital Zenica
Organization: Cantonal Hospital Zenica (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NR01/19
Record Dates: First submitted 2019-01-02; First posted 2019-01-04 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Insulin Resistance; Inflammatory Response; Exaggerated Well-Being; Length of Stay
Keywords: fasting; carbohydrate; insulin resistance
MeSH Terms: conditions — Insulin Resistance; Fasting

STUDY DESIGN:
Intervention Model Description: The diagnostic protocol for colon cancer was performed in patients at the surgery department. The patients with diagnosed colon tumor were prepared for the surgical procedure. After that, patients were examined to a preoperative anesthetic visit. During the visit, participants were assessed according to eligibility for enrollment in the study. The participants who have met the eligibility criteria have explained the nature of the study protocol. Those who agreed to participate in the study were randomized to one of two study groups for the duration of the study.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Surgeons, anesthetists, and outcome assessors were masking to the treatment allocation. Masking was possible because group allocation was performed by a nurse from the surgical ward, and the attending surgeon and anesthetist welcomed the participants at the operating room the next morning without knowledge of the type of intervention. The outcome study were evaluated by independent assessors who were also masked because they evaluated patients after surgery on a daily base during hospital stay without knowledge of the type intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAST group (No Intervention): preoperative fasting
- CHO group (Experimental): preoperative nutrition The participants of experimental group received 400 mil of a clear carbohydrate drink (12,5 gr/100 mil carbohydrate, 50 kcal/100ml, pH 5.0) at 10:00 pm the evening before surgery and another 200 mil of the carbohydrate drink on the day of surgery, 2 hours before induction of anesthesia. After surgery the participants fasted until the recovery of function of the bowel.
  Interventions: Dietary Supplement: preoperative nutrition

INTERVENTIONS:
Dietary Supplement: preoperative nutrition — The participants of experimental group received 400 mil of a clear carbohydrate drink (12,5 gr/100 mil carbohydrate, 50 kcal/100ml, pH 5.0) at 10:00 pm the evening before surgery and another 200 mil of the carbohydrate drink on the day of surgery, 2 hours before induction of anesthesia. After surgery the participants fasted until the recovery of function of the bowel.
  Arms: CHO group

SUMMARY:
This study compared traditional concept of preoperative fasting before elective open colon surgery and preoperative treatment with carbohydrate oral drink in intention to improve postoperative stress response to surgical procedure. Hypothesis was: preoperative oral carbohydrate drink reduces postoperative insulin resistance, improves insulin sensitivity, reduces postoperative inflammatory response in terms of the value of Glasgow Prognostic Score (GPS) and IL-6, improves postoperative patient's subjective well-being and surgical clinical outcome.

DETAILED DESCRIPTION:
This prospective randomized, controlled clinical study was carried out in the Department of Anesthesiology and Intensive Care Unit and Department of Surgery at the Cantonal Hospital Zenica, Bosnia and Herzegovina. After obtaining ethical committee approval 50 participants, scheduled for elective open colon surgery were included into study. Sample size was estimated using sample size calculator software and power analysis with 95% confidence interval and power of 80%. Statistical significance was considered as p< 0,05. The calculation indicated 19 participants per group would be sufficient to detect a 50% difference for insulin resistance between the groups. Assuming dropout would lead to a total sample size of 50 participants. Before each participant agreed to the join the study, the purpose and procedures of the study were fully explained and informed and written consent was obtained from each participant. A preoperative anesthetic examination was conducted the day before surgery. The participants who fulfilled study criteria were randomly allocated into two groups of 25 participants, depending on the preoperative treatment. The intervention group, received preoperative carbohydrate oral supplementation (CHO group) and the control group (FAST group) underwent to a conventional routine of preoperative fasting. Randomization was performed by computer generated randomization codes. The codes which indicated the treatment were held in sealed opaque envelopes. Nurse who conducted randomization and opened the envelopes the night before surgery was blinded to the study protocol as well as the surgeons, nurses, anesthesiologists and staff involved in data collection.

The participants of FAST group were undergone to the traditional concept of preoperative fasting before surgical procedure. The participants in the intervention group received carbohydrate oral supplement at 10:00 pm the evening before surgery and again on the day of surgery, 2 hours before induction of anesthesia. Assessment of clinical parameters started at 06:00 am on the day of surgery (basal value). The fasting peripheral venous blood samples were collected to measure serum levels of glucose, insulin, C-reactive protein, albumin and IL-6, and further 6 hours post-surgery, at 06.00 am on the first postoperative day and at 06:00 am on the second postoperative day. All patients underwent general anesthesia followed by colon surgery. Assessment of subjective well-being was performed immediately before induction into anesthesia using a 10 cm horizontal Visual Analogue Scales and then repeated for 0-4, 4-8, 8-12 and 12-24 hours post-surgery. Pain at rest, pain with mobilization, thirst, hunger, mouth dryness, anxiety and weakness were evaluated. The patients were explained how to use the scale. Surgical outcome was evaluated by postoperative return of gastrointestinal function, time to independent ambulation and postoperative discharge day. Postoperative data included and the time to oral intake. The following data were recorded also: age, sex, body weight, body mass index, American Society of Anesthesiologists (ASA) physical status class, nutritional status of the participants according to Nutritional Risk Screening 2002 (NRS-2002), tumor localization, type of surgery, duration of surgery, preoperative fasting time and, blood loss during surgery

ELIGIBILITY:
Inclusion Criteria:

* participants with ASA physical status class I-II
* aged between 18 years and 70 years
* participants scheduled for elective open colon surgery

Exclusion Criteria:

* previous treatment of colon or any other cancer
* disseminated malignant disease
* gastro-oesophageal reflux or increased risk of aspiration
* body mass index below 20 and above 30 kg/m2
* overall score ≥3 after final assessment of the nutritional status according to Nutritional Risk Screening 2002 (NRS-2002)
* emergency colon surgery
* diabetes mellitus
* inflammatory bowel disease
* immunological therapy
* cardiopulmonary disease
* neuromusular disease
* renal disease
* hepatic or endocrine disease
* pregnancy
* mental disease
* allergy to any study drugs
* alcoholic or drug abuse
* patient's refusal to participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-20 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
The mean change in insulin resistance using computer model Homeostasis model assessment of insulin resistance | blood samples were taken at 06:00 am on the day of surgery ( basal value), 6 hours post-surgery, at 06.00 am on the first postoperative day and at 06:00 am on the second postoperative day.
  Blood samples were collected to measure serum levels of glucose and serum levels of insulin. Insulin resistance, was calculated according to the equation = [fasting insulin (µU/ml) x fasting glucose (mmol/L)] / 22,5 using computer model Homeostasis model assessment of insulin resistance 2 Calculator version 2,2. The value >1 indicated the presence of resistance to insulin.
The mean change in Glasgow Prognostic Score (GPS). The GPS was obtained as ratio of serum C-reactive protein/albumin. | blood samples were taken at four time points: at 06:00 am on the day of surgery ( basal value), 6 hours post-surgery, at 06.00 am on the first postoperative day and at 06:00 am on the second postoperative day.
  The GPS was calculated as follow: participants with elevated level of C-reactive protein >10mg/L and albumin <35 g/L were allocated a score of 2. Participants showing one or neither of these blood chemistry abnormalities were allocated a score 1 or 0.
The mean change in serum level of IL-6 | blood samples were taken at four time points: at 06:00 am on the day of surgery ( basal value), 6 hours post-surgery, at 06.00 am on the first postoperative day and at 06:00 am on the second postoperative day.
  The concentration of IL-6 in serum has a r.n. 0-5,9 pg/mL.

SECONDARY OUTCOMES:
The mean change from baseline in participant's subjective well-being score on Visual Analogue Scale | The assessment of subjective well-being and pain score was performed immediately before induction into anesthesia and then repeated for 0-4, 4-8, 8-12 and 12-24 hours post-surgery
  The participant's subjective well-being included: pain at rest and with movement, thirst, hunger, dry mouth, weakness, anxiety, nausea and vomiting. The mean change were measured using a 10 cm horizontal Visual Analogue Scale. The scales were undivided and limited at both ends by vertical lines. The left end represented "no symptom" (score:0) and the right end represented "the worst imaginable" (score 100) limits of the variable to be evaluated. The participants rated discomfort by marking on the scales line at the point that represented their level of perceived symptom. The distance on the scales line from score 0 to the patient's mark determined the score of symptom intensity. The score was calculated as follow: 0-1cm no symptom; 1-3 cm mild symptom; 3-7 cm moderate symptom; 7-10 cm strong symptom. The patients were questioned about presence of nausea and vomiting at five study time points. A "NO" answer was grade as 1 and a "YES" answer was graded as 2.
surgical clinical outcomes | from 24 hours post-surgey from apprroximately 10 days post-surgery
  Surgical clinical outcomes included postoperative return of gastrointestinal function, time to independent ambulation and postoperative discharge day. The return of gastrointestinal function was assessed as follow: the sounds of the bowel were detected by an abdominal auscultation 24, 36, 48, 60, 72 and 80 hours after surgery. The time of the first postoperative flatus and defecation were recorded as well as the time to postoperative oral intake.

CONTACTS AND LOCATIONS:
Overall Officials: Nermina Rizvanović, MD, Principal Investigator — Cantonal Hospital Zenica, Crkvice 67, 72 000 Zenica, Bosnia and Herzegovina
Locations (1):
- Cantonal Hospital Zenica, Zenica, Bosnia and Herzegovina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Jodlowski T, Dobosz M. Preoperative fasting - is it really necessary? Pol Przegl Chir. 2014 Feb;86(2):100-5. doi: 10.2478/pjs-2014-0019. No abstract available. PMID 24670343
- [Result] Scott MJ, Baldini G, Fearon KC, Feldheiser A, Feldman LS, Gan TJ, Ljungqvist O, Lobo DN, Rockall TA, Schricker T, Carli F. Enhanced Recovery After Surgery (ERAS) for gastrointestinal surgery, part 1: pathophysiological considerations. Acta Anaesthesiol Scand. 2015 Nov;59(10):1212-31. doi: 10.1111/aas.12601. Epub 2015 Sep 8. PMID 26346577
- [Result] Ljungqvist O. Jonathan E. Rhoads lecture 2011: Insulin resistance and enhanced recovery after surgery. JPEN J Parenter Enteral Nutr. 2012 Jul;36(4):389-98. doi: 10.1177/0148607112445580. Epub 2012 May 10. PMID 22577121
- [Result] Akbarzadeh M, Eftekhari MH, Shafa M, Alipour S, Hassanzadeh J. Effects of a New Metabolic Conditioning Supplement on Perioperative Metabolic Stress and Clinical Outcomes: A Randomized, Placebo-Controlled Trial. Iran Red Crescent Med J. 2016 Jan 9;18(1):e26207. doi: 10.5812/ircmj.26207. eCollection 2016 Jan. PMID 26889394
- [Result] Witasp A, Nordfors L, Schalling M, Nygren J, Ljungqvist O, Thorell A. Expression of inflammatory and insulin signaling genes in adipose tissue in response to elective surgery. J Clin Endocrinol Metab. 2010 Jul;95(7):3460-9. doi: 10.1210/jc.2009-2588. Epub 2010 May 5. PMID 20444921
- [Result] Costa MD, Vieira de Melo CY, Amorim AC, Cipriano Torres Dde O, Dos Santos AC. Association Between Nutritional Status, Inflammatory Condition, and Prognostic Indexes with Postoperative Complications and Clinical Outcome of Patients with Gastrointestinal Neoplasia. Nutr Cancer. 2016 Oct;68(7):1108-14. doi: 10.1080/01635581.2016.1206578. Epub 2016 Aug 2. PMID 27485861
- [Result] Gomes de Lima KV, Maio R. Nutritional status, systemic inflammation and prognosis of patients with gastrointestinal cancer. Nutr Hosp. 2012 May-Jun;27(3):707-14. doi: 10.3305/nh/2012.27.3.5567. PMID 23114934
- [Result] Ishizuka M, Nagata H, Takagi K, Iwasaki Y, Shibuya N, Kubota K. Clinical Significance of the C-Reactive Protein to Albumin Ratio for Survival After Surgery for Colorectal Cancer. Ann Surg Oncol. 2016 Mar;23(3):900-7. doi: 10.1245/s10434-015-4948-7. Epub 2015 Nov 3. PMID 26530445
- [Result] Perrone F, da-Silva-Filho AC, Adorno IF, Anabuki NT, Leal FS, Colombo T, da Silva BD, Dock-Nascimento DB, Damiao A, de Aguilar-Nascimento JE. Effects of preoperative feeding with a whey protein plus carbohydrate drink on the acute phase response and insulin resistance. A randomized trial. Nutr J. 2011 Jun 13;10:66. doi: 10.1186/1475-2891-10-66. PMID 21668975
- [Result] Nygren J. The metabolic effects of fasting and surgery. Best Pract Res Clin Anaesthesiol. 2006 Sep;20(3):429-38. doi: 10.1016/j.bpa.2006.02.004. PMID 17080694
- [Result] Kratzing C. Pre-operative nutrition and carbohydrate loading. Proc Nutr Soc. 2011 Aug;70(3):311-5. doi: 10.1017/S0029665111000450. PMID 21781358
- [Result] Sada F, Krasniqi A, Hamza A, Gecaj-Gashi A, Bicaj B, Kavaja F. A randomized trial of preoperative oral carbohydrates in abdominal surgery. BMC Anesthesiol. 2014 Oct 17;14:93. doi: 10.1186/1471-2253-14-93. eCollection 2014. PMID 25364300
- [Result] Gianotti L, Biffi R, Sandini M, Marrelli D, Vignali A, Caccialanza R, Vigano J, Sabbatini A, Di Mare G, Alessiani M, Antomarchi F, Valsecchi MG, Bernasconi DP. Preoperative Oral Carbohydrate Load Versus Placebo in Major Elective Abdominal Surgery (PROCY): A Randomized, Placebo-controlled, Multicenter, Phase III Trial. Ann Surg. 2018 Apr;267(4):623-630. doi: 10.1097/SLA.0000000000002325. PMID 28582271
- [Result] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Result] Amer MA, Smith MD, Herbison GP, Plank LD, McCall JL. Network meta-analysis of the effect of preoperative carbohydrate loading on recovery after elective surgery. Br J Surg. 2017 Feb;104(3):187-197. doi: 10.1002/bjs.10408. Epub 2016 Dec 21. PMID 28000931
- [Result] Sarin A, Chen LL, Wick EC. Enhanced recovery after surgery-Preoperative fasting and glucose loading-A review. J Surg Oncol. 2017 Oct;116(5):578-582. doi: 10.1002/jso.24810. Epub 2017 Aug 28. PMID 28846137
- [Result] Smith MD, McCall J, Plank L, Herbison GP, Soop M, Nygren J. Preoperative carbohydrate treatment for enhancing recovery after elective surgery. Cochrane Database Syst Rev. 2014 Aug 14;2014(8):CD009161. doi: 10.1002/14651858.CD009161.pub2. PMID 25121931
- [Result] Kang ZQ, Huo JL, Zhai XJ. Effects of perioperative tight glycemic control on postoperative outcomes: a meta-analysis. Endocr Connect. 2018 Dec 1;7(12):R316-R327. doi: 10.1530/EC-18-0231. PMID 30120204
- [Result] Gillis C, Carli F. Promoting Perioperative Metabolic and Nutritional Care. Anesthesiology. 2015 Dec;123(6):1455-72. doi: 10.1097/ALN.0000000000000795. PMID 26248016
- [Result] Pinto Ados S, Grigoletti SS, Marcadenti A. Fasting abbreviation among patients submitted to oncologic surgery: systematic review. Arq Bras Cir Dig. 2015;28(1):70-3. doi: 10.1590/S0102-67202015000100018. PMID 25861075
- [Result] Tamura T, Yatabe T, Kitagawa H, Yamashita K, Hanazaki K, Yokoyama M. Oral carbohydrate loading with 18% carbohydrate beverage alleviates insulin resistance. Asia Pac J Clin Nutr. 2013;22(1):48-53. doi: 10.6133/apjcn.2013.22.1.20. PMID 23353610
- [Result] Pexe-Machado PA, de Oliveira BD, Dock-Nascimento DB, de Aguilar-Nascimento JE. Shrinking preoperative fast time with maltodextrin and protein hydrolysate in gastrointestinal resections due to cancer. Nutrition. 2013 Jul-Aug;29(7-8):1054-9. doi: 10.1016/j.nut.2013.02.003. PMID 23759267
- [Result] Feng J, Li K, Li L, Wang X, Huang M, Yang J, Hu Y. The effects of fast-track surgery on inflammation and immunity in patients undergoing colorectal surgery. Int J Colorectal Dis. 2016 Oct;31(10):1675-82. doi: 10.1007/s00384-016-2630-6. Epub 2016 Aug 12. PMID 27517680
- [Result] Barbic J, Ivic D, Alkhamis T, Drenjancevic D, Ivic J, Harsanji-Drenjancevic I, Turina I, Vcev A. Kinetics of changes in serum concentrations of procalcitonin, interleukin-6, and C- reactive protein after elective abdominal surgery. Can it be used to detect postoperative complications? Coll Antropol. 2013 Mar;37(1):195-201. PMID 23697273
- [Result] Weimann A, Braga M, Carli F, Higashiguchi T, Hubner M, Klek S, Laviano A, Ljungqvist O, Lobo DN, Martindale R, Waitzberg DL, Bischoff SC, Singer P. ESPEN guideline: Clinical nutrition in surgery. Clin Nutr. 2017 Jun;36(3):623-650. doi: 10.1016/j.clnu.2017.02.013. Epub 2017 Mar 7. PMID 28385477
- [Result] Kadoi Y. Blood glucose control in the perioperative period. Minerva Anestesiol. 2012 May;78(5):574-95. Epub 2012 Feb 10. PMID 22327042
- [Result] Hausel J, Nygren J, Lagerkranser M, Hellstrom PM, Hammarqvist F, Almstrom C, Lindh A, Thorell A, Ljungqvist O. A carbohydrate-rich drink reduces preoperative discomfort in elective surgery patients. Anesth Analg. 2001 Nov;93(5):1344-50. doi: 10.1097/00000539-200111000-00063. PMID 11682427
- [Result] Burgess LC, Phillips SM, Wainwright TW. What Is the Role of Nutritional Supplements in Support of Total Hip Replacement and Total Knee Replacement Surgeries? A Systematic Review. Nutrients. 2018 Jun 25;10(7):820. doi: 10.3390/nu10070820. PMID 29941852
- [Result] Awad S, Varadhan KK, Ljungqvist O, Lobo DN. A meta-analysis of randomised controlled trials on preoperative oral carbohydrate treatment in elective surgery. Clin Nutr. 2013 Feb;32(1):34-44. doi: 10.1016/j.clnu.2012.10.011. Epub 2012 Nov 7. PMID 23200124